CLINICAL TRIAL: NCT02027532
Title: Prevention of Infection in Surgical Treatment of Closed Fractures: A Comparative Study of Cefazolin Versus Vancomycin
Brief Title: Prevention of Infection in Closed Fractures: Cefazolin Versus Vancomycin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not complete study due to administrative challenges
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09-060; NCT01029457 (obsolete NCT alias)
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2017-05

CONDITIONS: Infection; Closed Fractures
MeSH Terms: conditions — Infections; Fractures, Closed | interventions — Cefazolin; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Active Comparator): intravenous, weight-based dose (1gm<80kg, 2gm>80kg), perioperatively
  Interventions: Drug: Cefazolin
- Vancomycin (Active Comparator): intravenous, weight-based dose (1gm<80kg, 2gm>80kg), perioperatively
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Cefazolin
  Arms: Cefazolin
Drug: Vancomycin
  Arms: Vancomycin

SUMMARY:
The purpose of this study is to compare the incidence rate of infection in surgical patients with closed fractures treated prophylactically with Cefazolin versus Vancomycin in the peri-operative period.

The hypothesis of this study is that patients undergoing surgical treatment for closed fractures who are treated prophylactically with Vancomycin will have a lower incidence rate of infection than patients who are treated prophylactically with Cefazolin.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 years old and 85 years old
* Closed fracture
* Fracture treatment plan is for one operation on one day (one surgical setting)
* Likely to follow-up with surgeon until fracture is healed
* Ability to understand and agree to Informed Consent

Exclusion Criteria:

* Under 18 years old or over 85 years old
* Open fracture(s)
* Fracture requires multiple operations
* Other injuries requiring operations
* Documented allergy to Cefazolin or Vancomycin
* Previous history of Methicillin-resistant Staphylococcus aureus infection
* Previous surgery on the injured extremity within 1 year
* Use of antibiotics within 2 weeks before or after injury
* Use of antibiotics within 2 weeks before surgery
* Unlikely to follow-up until fracture is healed
* Unable to understand and agree to Informed Consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2009-10; Primary Completion 2015-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
incidence of infection | one year

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Nowotarski, M.D., Principal Investigator — UTCOM Chattanooga/Erlanger Health System
Locations (1):
- Erlanger Health System, Chattanooga, Tennessee, United States